CLINICAL TRIAL: NCT00717769
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Study of SUN13834 in Adult Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASBI 404
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; SUN13834
MeSH Terms: conditions — Dermatitis, Atopic | interventions — 6-(5-chloro-2-methoxybenzyl)-4-alarkylaminocarbonyl-1,4-diazepane-2,5-dione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SUN13834 (Experimental)
  Interventions: Drug: SUN13834
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SUN13834 — Low dose, orally 3 times a day (tid) for 28 days of SUN13834
  Arms: SUN13834
Drug: Placebo — Placebo, orally (tid) for 28 days of SUN13834
  Arms: Placebo

SUMMARY:
The purpose of the study is to explore the efficacy and safety of SUN13834 vs placebo in adult participants with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 18 and 65 years of age.
* A diagnosis of Atopic Dermatitis (AD), meeting the Guidelines for Diagnosis of Atopic Dermatitis criteria
* At least 1 inflammatory lesion Eczema Area and Severity Index (EASI) score ≥5 at Screening and prior to randomization (as per Amendment 2 and 3). Under the original protocol and Amendment 1, no minimum EASI score was required.

Exclusion Criteria:

* Taking systemic immunosuppressive drugs or biologicals (within 3 months), or systemic corticosteroids therapy (within 4 weeks)prior to Screening(note: inhaled, intranasal or otic corticosteroids are allowed).
* Use of phototherapy or tanning beds within 6 weeks of screening
* History of reactive airway disease (asthma) requiring hospitalization in an intensive care unit in the last 5 years.
* Presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the Clinical Investigator) that will interfere with the interpretation of data from this patient (eg, renal impairment with non-atopic pruritus).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2008-07-16 (Actual); Primary Completion 2009-04-09 (Actual); Study Completion 2009-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (28):
- United States (28):
  - Radiant Research, Inc., Birmingham, Alabama
  - Pivotal Research Center, Mesa, Arizona
  - Pivotal Research Center, Peoria, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Therapeutics Clinical Research, San Diego, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Miami Research Associates, Miami, Florida
  - Advanced Dermatology and Cosmetic Surgery, Ormond Beach, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - Deaconess Clinic Downtown Research Institute, Evansville, Indiana
  - DermResearch, PLLC, Louisville, Kentucky
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Academic Dermatology, Albuquerque, New Mexico
  - Derm Research Center of New York, Inc., Stony Brook, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Wake Forest University Health Sciences - Dermatology Studies, Winston-Salem, North Carolina
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Oklahoma University Health Sciences Center, Dermatology Dept, Oklahoma City, Oklahoma
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Radiant Research, Inc, Greer, South Carolina
  - J & S Studies, Inc, College Station, Texas
  - Baylor Research Institute of Dermatology Department, Dallas, Texas
  - Dermatology Associates of San Antonio, San Antonio, Texas
  - Intermountain Clinical Research, Draper, Utah
  - Commonwealth Clinical Research Specialists, Inc., Richmond, Virginia
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 270 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 27 clinic sites in the United States of America (USA).
Pre-assignment Details: Washout period for Atopic Dermatitis treatments such as topical corticosteroids, antihistamines, over the counter (OTC) sleep aids, and some FDA approved devices for 3 months up to 1 week prior to screening and for the duration of the study (including follow-up). After the initiation of the study, the protocol was amended to discontinue group 3 (200 mg three times a day [tid]). The efficacy outcomes and analyses were also redefined to compare the 50 mg tid group against the placebo group.
Groups:
- Placebo: Participants with atopic dermatitis who were administered 2 SUN13834-matching placebo tablets orally 3 times a day (tid) for 28 days.
- SUN13834 50 mg Tid: Participants with atopic dermatitis who were administered 2 SUN13834 tablets of 25 mg; 50 mg (2×25 mg) orally tid for 28 days.
- SUN13834 200 mg Tid: Participants with atopic dermatitis who were administered 2 SUN13834 tablets of 100 mg; 200 mg (2×100 mg) orally tid for 28 days.
Period: Overall Study
Arm/Group | Placebo | SUN13834 50 mg Tid | SUN13834 200 mg Tid
Started | 120 | 120 | 30
Completed | 104 | 102 | 19
Not Completed | 16 | 18 | 11
Not completed — Adverse Event | 9 | 6 | 1
Not completed — Lack of compliance | 0 | 2 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Sponsor decision | 1 | 0 | 10
Not completed — Withdrew consent | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Intent-to-treat (ITT) population.
Groups:
- SUN13834 50 mg Tid: Participants with atopic dermatitis who were administered 2 SUN13834 tablets of 25 mg;(2×50 mg) orally tid for 28 days.
- SUN13834 200 mg Tid: Participants with atopic dermatitis who were administered 2 SUN13834 tablets of 200 mg (2×100 mg) orally tid for 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | SUN13834 50 mg Tid | SUN13834 200 mg Tid | Total
Number analyzed (Participants) | 120 | 119 | 30 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (13.14) | 38.5 (12.95) | 37.0 (10.62) | 37.8 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 60 | 22 | 154
  Male | 48 | 59 | 8 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 0 | 23
  Not Hispanic or Latino | 109 | 107 | 30 | 246
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 46 | 50 | 9 | 105
  White | 71 | 65 | 21 | 157
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 120 | 119 | 30 | 269

OUTCOME MEASURES:

1. Primary Outcome: Baseline of Disease Characteristics Before Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: Eczema Area and Severity Index (EASI) Score is a composite index including an assessment of disease extent and percent of body surface area involved, converted to a proportional factor in 4 body regions (head and neck, lower limbs, upper limbs, and trunk). The total EASI has a minimum score of 0 (clear) and a maximum of 72 (very severe). Investigator's Global Assessment (IGA) score consists of a 6-point scale from a minimum of 0 (clear) and a maximum of 6 (very severe atopic dermatitis). (0 = clear; 1 = almost clear; 2 = mild disease; 3 = moderate disease, 4 = severe disease; and 5 = very severe disease). Pruritus score consists of a 4-point scale with 0 as the minimum and 3 as the maximum (0 = absent, 1 = mild, 2 = moderate, 3 = severe). Insomnia score is an 11-point scale, ranging from a minimum of no insomnia (score = 0) to a maximum of severe insomnia (score = 10). Higher scores indicate a worse outcome and lower scores indicate a better outcome for all scales.
Time Frame: Pre-dose
Population: Baseline disease characteristics were assessed using the Intent-to-Treat (ITT) population. All enrolled participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid | SUN13834 200 mg Tid
Number analyzed (Participants) | 120 | 119 | 30
score on a scale
  Eczema Area and Severity Index (EASI) Score | 12.59 (10.02) | 12.45 (8.75) | 6.01 (5.98)
  Investigator's Global Assessment (IGA) Score | 3.0 (0.67) | 3.1 (0.69) | 2.6 (0.93)
  Pruritus Score | 2.2 (0.74) | 2.2 (0.72) | 1.9 (0.80)
  Insomnia Score | 3.2 (3.16) | 4.0 (3.06) | 3.0 (3.07)

2. Primary Outcome: Mean Change in Eczema Area and Severity Index (EASI) Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: EASI is an overall assessment of the disease severity of the entire body. The EASI is a composite index including an assessment of disease extent and percent of body surface area involved, converted to a proportional factor (scale of 0-6), in 4 body regions (head and neck, lower limbs, upper limbs, and trunk). The EASI also includes an assessment of erythema, induration and/or papulation, excoriation, and lichenification, each on a scale of 0 to 3. The EASI has a minimum score of 0 (clear) and a maximum of 72 (very severe). The algorithm for calculating the EASI requires, for each body region, the sum of the clinical sign scores multiplied by the area, multiplied by the proportional factor. The total EASI score is the sum of the 4 body region scores. A negative value is an indication of a decrease in individual EASI scores and eczema severity. Higher scores indicate a worse outcome and lower scores a better outcome.
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: EASI score was assessed using the Intent-to-Treat population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 120 | 119
units on a scale
  Day 8: Change from Baseline | -1.66 (4.59) | -1.94 (3.36)
  Day 15: Change from Baseline | -2.88 (4.82) | -4.06 (4.92)
  Day 22: Change from Baseline | -3.83 (6.30) | -5.67 (6.60)
  Day 29: Change from Baseline | -4.70 (6.96) | -6.70 (6.82)
  Follow-up Week 2: Change from Baseline | -4.64 (6.70) | -6.41 (7.86)
  Follow-up Week 4: Change from Baseline | -4.41 (6.95) | -6.73 (7.77)
Statistical Analysis 1: Comparison: Placebo vs SUN13834 50 mg Tid; Change from Baseline to Day 8; Test type: Superiority; p = 0.519, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs SUN13834 50 mg Tid; Change from Baseline to Day 15; Test type: Superiority; p = 0.032, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs SUN13834 50 mg Tid; Change from Baseline to Day 22; Test type: Superiority; p = 0.008, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs SUN13834 50 mg Tid; Change from Baseline to Day 29; Test type: Superiority; p = 0.006, ANCOVA

3. Primary Outcome: Percent Change in Eczema Area and Severity Index (EASI) Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 2
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 120 | 119
percent change
  Day 8: % Change from Baseline | -12.62 (30.45) | -15.52 (27.03)
  Day 15: % Change from Baseline | -23.42 (33.34) | -28.46 (59.41)
  Day 22: % Change from Baseline | -30.83 (42.61) | -39.11 (42.83)
  Day 29: % Change from Baseline | -38.33 (43.89) | -47.46 (39.89)
  Follow-up Week 2: % Change from Baseline | -37.29 (56.64) | -45.35 (45.55)
  Follow-up Week 4: % Change from Baseline | -37.89 (53.35) | -48.06 (44.46)

4. Primary Outcome: Mean Change in Eczema Area and Severity Index (EASI) Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 2
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: EASI was assessed from the Efficacy Evaluable population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 93 | 87
units on a scale
  Day 8: Change from Baseline | -1.94 (5.08) | -2.36 (3.73)
  Day 15: Change from Baseline | -3.28 (5.27) | -5.13 (4.95)
  Day 22: Change from Baseline | -4.26 (6.91) | -7.08 (6.81)
  Day 29: Change from Baseline | -5.26 (7.55) | -8.19 (6.90)
  Follow-up Week 2: Change from Baseline | -5.38 (7.20) | -7.99 (8.29)
  Follow-up Week 4: Change from Baseline | -5.09 (7.24) | -8.49 (7.89)
Statistical Analysis 1: Comparison: Placebo vs SUN13834 50 mg Tid; Change from Baseline to Day 8; Test type: Superiority; p = 0.533, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs SUN13834 50 mg Tid; Change from Baseline to Day 15; Test type: Superiority; p = 0.009, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs SUN13834 50 mg Tid; Change from Baseline to Day 22; Test type: Superiority; p = 0.002, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs SUN13834 50 mg Tid; Change from Baseline to Day 29; Test type: Superiority; p = 0.003, ANCOVA

5. Primary Outcome: Percent Change in Eczema Area and Severity Index (EASI) Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 2
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: EASI score was assessed using the Efficacy Evaluable population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 93 | 87
percent change
  Day 8: % Change from Baseline | -13.65 (29.51) | -16.03 (23.94)
  Day 15: % Change from Baseline | -23.67 (31.94) | -33.64 (31.26)
  Day 22: % Change from Baseline | -29.29 (45.21) | -44.40 (35.29)
  Day 29: % Change from Baseline | -37.58 (46.18) | -52.84 (35.90)
  Follow-up Week 2: % Change from Baseline | -40.69 (46.07) | -50.86 (42.50)
  Follow-up Week 4: % Change from Baseline | -40.16 (47.42) | -54.35 (40.40)

6. Secondary Outcome: Mean Change in Investigator's Global Assessment (IGA) Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: IGA score is used as an overall assessment of disease severity of the entire body, which consists of a 6-point scale from a minimum of 0 (clear) and a maximum of 6 (very severe atopic dermatitis). Higher scores indicate a worse outcome and lower scores indicate a better outcome. (0 = clear; 1 = almost clear; 2 = mild disease; 3 = moderate disease, 4 = severe disease; and 5 = very severe disease).
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: IGA Score was assessed from the Intent-To-Treat population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 120 | 119
units on a scale
  Day 8: Change from Baseline | -0.2 (0.54) | -0.3 (0.57)
  Day 15: Change from Baseline | -0.4 (0.69) | -0.6 (0.74)
  Day 22: Change from Baseline | -0.6 (0.77) | -0.9 (0.87)
  Day 29: Change from Baseline | -0.8 (0.97) | -1.1 (1.00)
  Follow-up Week 2: Change from Baseline | -0.8 (1.01) | -1.1 (1.05)
  Follow-up Week 4: Change from Baseline | -0.8 (1.10) | -1.1 (1.04)

7. Secondary Outcome: Percent Change in Investigator's Global Assessment (IGA) Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 6
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 120 | 119
percent change
  Day 8: % Change from Baseline | -6.10 (18.51) | -8.83 (18.17)
  Day 15: % Change from Baseline | -10.84 (23.00) | -19.99 (32.34)
  Day 22: % Change from Baseline | -17.95 (26.13) | -28.89 (30.57)
  Day 29: % Change from Baseline | -24.21 (32.24) | -34.93 (34.42)
  Follow-up Week 2: % Change from Baseline | -25.91 (34.47) | -34.48 (36.66)
  Follow-up Week 4: % Change from Baseline | -27.24 (37.59) | -34.10 (36.67)

8. Secondary Outcome: Mean Change in Investigator's Global Assessment (IGA) Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 6
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: IGA Score was assessed from the Efficacy Evaluable population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 93 | 87
units on a scale
  Day 8: Change from Baseline | -0.2 (0.54) | -0.2 (0.58)
  Day 15: Change from Baseline | -0.4 (0.66) | -0.7 (0.69)
  Day 22: Change from Baseline | -0.5 (0.80) | -1.0 (0.83)
  Day 29: Change from Baseline | -0.8 (1.02) | -1.2 (0.98)
  Follow-up Week 2: Change from Baseline | -0.8 (1.05) | -1.2 (1.04)
  Follow-up Week 4: Change from Baseline | -0.8 (1.13) | -1.2 (1.05)

9. Secondary Outcome: Percent Change in Investigator's Global Assessment (IGA) Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 6
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 93 | 87
percent change
  Day 8: % Change from Baseline | -7.06 (17.76) | -7.33 (17.38)
  Day 15: % Change from Baseline | -11.09 (21.72) | -20.23 (20.93)
  Day 22: % Change from Baseline | -16.02 (26.71) | -30.47 (24.68)
  Day 29: % Change from Baseline | -23.64 (33.88) | -37.99 (29.96)
  Follow-up Week 2: % Change from Baseline | -25.18 (35.21) | -36.51 (32.98)
  Follow-up Week 4: % Change from Baseline | -25.72 (37.31) | -37.43 (34.26)

10. Secondary Outcome: Mean Change in Pruritus Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: Symptoms of pruritus were assessed using the Pruritus score. The Pruritus score consists of a 4-point scale with 0 as the minimum and 3 as the maximum (0 = absent, 1 = mild, 2 = moderate, 3 = severe). A lower score (0) indicates a better outcome and a higher score (3) indicates a worse outcome. A negative value indicates a decreasing change in the pruritus score. A negative value is an indication of a decrease in individual scores.
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: Pruritus score was assessed from the Intent-To-Treat population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 120 | 119
units on a scale
  Day 8: Change from Baseline | -0.3 (0.77) | -0.3 (0.88)
  Day 15: Change from Baseline | -0.5 (0.83) | -0.6 (0.92)
  Day 22: Change from Baseline | -0.6 (0.92) | -0.7 (1.04)
  Day 29: Change from Baseline | -0.7 (0.85) | -0.9 (1.04)
  Follow-up Week 2: Change from Baseline | -0.6 (1.04) | -0.8 (1.09)
  Follow-up Week 4: Change from Baseline | -0.6 (0.93) | -0.7 (1.09)

11. Secondary Outcome: Percent Change in Pruritus Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 10
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 120 | 119
percent change
  Day 8: % Change from Baseline | -1.54 (99.05) | -7.68 (48.73)
  Day 15: % Change from Baseline | -11.53 (101.25) | -22.22 (48.74)
  Day 22: % Change from Baseline | -13.89 (104.86) | -25.99 (54.76)
  Day 29: % Change from Baseline | -18.75 (103.37) | -33.34 (51.94)
  Follow-up Week 2: % Change from Baseline | -11.95 (109.12) | -28.11 (55.80)
  Follow-up Week 4: % Change from Baseline | -15.14 (106.67) | -27.82 (53.91)

12. Secondary Outcome: Mean Change in Pruritus Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 10
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: Pruritus score was assessed from the Efficacy Evaluable population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 93 | 87
units on a scale
  Day 8: Change from Baseline | -0.3 (0.72) | -0.3 (0.87)
  Day 15: Change from Baseline | -0.5 (0.80) | -0.7 (0.95)
  Day 22: Change from Baseline | -0.6 (0.91) | -0.7 (1.10)
  Day 29: Change from Baseline | -0.7 (0.89) | -0.9 (1.13)
  Follow-up Week 2: Change from Baseline | -0.6 (1.06) | -0.7 (1.16)
  Follow-up Week 4: Change from Baseline | -0.6 (0.91) | -0.7 (1.14)

13. Secondary Outcome: Percent Change in Pruritus Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 10
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 93 | 87
percent change
  Day 8: % Change in Baseline | -10.03 (31.19) | -7.45 (44.81)
  Day 15: % Change from Baseline | -17.92 (38.01) | -23.45 (50.45)
  Day 22: % Change from Baseline | -20.25 (44.70) | -22.61 (57.74)
  Day 29: % Change from Baseline | -24.73 (45.75) | -33.34 (56.78)
  Follow-up Week 2: % Change from Baseline | -21.69 (55.60) | -24.72 (57.34)
  Follow-up Week 4: % Change from Baseline | -22.76 (46.81) | -22.41 (54.15)

14. Secondary Outcome: Mean Change in Insomnia Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: The extent of insomnia experienced by the participant was assessed using the Insomnia score. The Insomnia score is an 11-point scale, ranging from a minimum of no insomnia (score = 0) to a maximum of severe insomnia (score = 10). A lower score (0) indicates a better outcome and a higher score (10) indicates a worse outcome. A negative value indicates a decreasing change in the insomnia score. A negative value is an indication of a decrease in individual scores.
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: Insomnia score was assessed from the Intent-To-Treat population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 120 | 119
units on a scale
  Day 8: Change from Baseline | -0.6 (2.50) | -0.7 (2.61)
  Day 15: Change from Baseline | -0.7 (2.50) | -1.2 (2.69)
  Day 22: Change from Baseline | -0.8 (2.48) | -1.3 (2.96)
  Day 29: Change from Baseline | -0.9 (2.55) | -1.4 (3.01)
  Follow-up Week 2: Change from Baseline | -0.9 (2.77) | -1.1 (3.12)
  Follow-up Week 4: Change from Baseline | -0.8 (2.88) | -1.3 (3.24)

15. Secondary Outcome: Mean Change in Insomnia Score From Baseline to Each Visit Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: as for outcome 14
Time Frame: Day 8, Day 15, Day 22, Day 29, Follow Up Week 2 and Week 4 post-dose.
Population: Insomnia score was assessed from the Efficacy Evaluable population. Based on the emended protocol, 50 mg tid and the placebo groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN13834 50 mg Tid
Number analyzed (Participants) | 93 | 87
units on a scale
  Day 8: Change from Baseline | -0.6 (2.41) | -0.7 (2.78)
  Day 15: Change from Baseline | -0.7 (2.20) | -1.3 (2.66)
  Day 22: Change from Baseline | -0.6 (2.25) | -1.4 (2.93)
  Day 29: Change from Baseline | -0.8 (2.44) | -1.5 (2.96)
  Follow-up Week 2: Change from Baseline | -0.9 (2.50) | -1.0 (3.09)
  Follow-up Week 4: Change from Baseline | -0.6 (2.56) | -1.3 (3.17)

16. Secondary Outcome: Mean of SUN13834 Plasma Concentrations Over Time Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Time Frame: Baseline up to 0-2.5 h, 2.5-5.0 h, 5.0-10 h, 8-24 h post-dose.
Population: Mean of SUN13834 Plasma Concentrations were assessed from the Pharmacokinetic-Intent-to-Treat (PK-ITT) population, those with evaluable data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SUN13834 50 mg Tid | SUN13834 200 mg Tid
Number analyzed (Participants) | 107 | 27
ng/mL
  Predose | 0.565 (4.81) | 0.100 (NA) — Mean plasma SUN13834 at pre-dose for the PK-ITT population is <0.100. Below the level of detection.
  0-2.5 h: number analyzed (Participants) | 105 | 25
  0-2.5 h | 99.8 (119) | 452 (691)
  2.5-5.0 h: number analyzed (Participants) | 98 | 17
  2.5-5.0 h | 90.6 (86.7) | 367 (237)
  5.0-10 h: number analyzed (Participants) | 91 | 22
  5.0-10 h | 49.4 (69.8) | 120 (122)
  8-24 h: number analyzed (Participants) | 71 | 11
  8-24 h | 27.2 (98.1) | 29.2 (34.0)

17. Secondary Outcome: Mean of SUN13834 Plasma Concentrations Over Time Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Time Frame: Baseline up to 0-2.5 h, 2.5-5.0 h, 5.0-10 h, 8-24 h post-dose.
Population: Mean of SUN13834 Plasma Concentrations were assessed from the Pharmacokinetic-Efficacy Evaluable (PK-EE) population, those with evaluable data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SUN13834 50 mg Tid | SUN13834 200 mg Tid
Number analyzed (Participants) | 77 | 8
ng/mL
  Predose | 0.747 (5.68) | 0.100 (NA) — Mean plasma SUN13834 at pre-dose for the PK-EE population is <0.100. Below level of detection.
  0-2.5 h: number analyzed (Participants) | 77 | 7
  0-2.5 h | 93.7 (122) | 741 (1090)
  2.5-5.0 h: number analyzed (Participants) | 75 | 6
  2.5-5.0 h | 87.7 (86.7) | 508 (270)
  5.0-10 h: number analyzed (Participants) | 70 | 6
  5.0-10 h | 50.5 (78.5) | 103 (76.4)
  8-24 h: number analyzed (Participants) | 61 | 3
  8-24 h | 18.2 (51.7) | 11.3 (4.47)

18. Secondary Outcome: Mean of SUN13834 Metabolite Plasma Concentrations Over Time Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: Mean concentrations of SUN13834 metabolites M-3, M-5, M-6, M-6G, MG-1, and MG-2 in participant plasma samples were measured.
Time Frame: Baseline up to 0-2.5 h, 2.5-5.0 h, 5.0-10 h, 8-24 h post-dose.
Population: Mean of SUN13834 metabolite plasma concentrations were assessed using the Pharmacokinetic-Intent-to-Treat (PK-ITT) population, those with evaluable data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SUN13834 50 mg Tid | SUN13834 200 mg Tid
Number analyzed (Participants) | 107 | 27
ng/mL
  M-3: Predose | 0.500 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is <0.500. Below level of detection. | 0.500 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is <0.500. Below level of detection.
  M-3: 0-2.5 h: number analyzed (Participants) | 105 | 25
  M-3: 0-2.5 h | 7.59 (8.77) | 32.9 (48.4)
  M-3: 2.5-5.0 h: number analyzed (Participants) | 98 | 17
  M-3: 2.5-5.0 h | 8.01 (6.27) | 41.7 (28.4)
  M-3:5.0-10 h: number analyzed (Participants) | 91 | 22
  M-3:5.0-10 h | 4.36 (5.10) | 13.2 (14.4)
  M-3: 8-24 h: number analyzed (Participants) | 71 | 11
  M-3: 8-24 h | 2.33 (6.79) | 6.11 (10.0)
  M-5: Predose | 0.513 (0.132) | 0.500 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is <0.500. Below level of detection.
  M-5: 0-2.5 h: number analyzed (Participants) | 105 | 25
  M-5: 0-2.5 h | 16.8 (17.3) | 76.9 (122)
  M-5: 2.5-5.0 h: number analyzed (Participants) | 98 | 17
  M-5: 2.5-5.0 h | 17.0 (13.0) | 68.1 (70.9)
  M-5:5.0-10 h: number analyzed (Participants) | 91 | 22
  M-5:5.0-10 h | 13.0 (11.7) | 33.3 (19.6)
  M-5: 8-24 h: number analyzed (Participants) | 71 | 11
  M-5: 8-24 h | 8.91 (18.0) | 16.8 (17.4)
  M-6: Predose | 0.500 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is <0.500. Below level of detection. | 0.500 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is <0.500. Below level of detection.
  M-6: 0-2.5 h: number analyzed (Participants) | 105 | 25
  M-6: 0-2.5 h | 26.8 (26.8) | 69.5 (83.7)
  M-6: 2.5-5.0 h: number analyzed (Participants) | 98 | 17
  M-6: 2.5-5.0 h | 31.6 (21.5) | 96.6 (67.4)
  M-6:5.0-10 h: number analyzed (Participants) | 91 | 22
  M-6:5.0-10 h | 26.6 (19.6) | 65.7 (50.9)
  M-6: 8-24 h: number analyzed (Participants) | 71 | 11
  M-6: 8-24 h | 16.9 (43.8) | 50.0 (79.1)
  M-6G: Predose | 0.00 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is 0. Below level of detection. | 0.00 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is 0. Below level of detection.
  M-6G: 0-2.5 h: number analyzed (Participants) | 105 | 25
  M-6G: 0-2.5 h | 15.3 (22.8) | 26.1 (41.3)
  M-6G: 2.5-5.0 h: number analyzed (Participants) | 98 | 17
  M-6G: 2.5-5.0 h | 18.9 (22.3) | 85.3 (63.6)
  M-6G:5.0-10 h: number analyzed (Participants) | 91 | 22
  M-6G:5.0-10 h | 16.2 (17.9) | 54.4 (61.8)
  M-6G: 8-24 h: number analyzed (Participants) | 71 | 11
  M-6G: 8-24 h | 12.6 (25.7) | 34.1 (55.1)
  MG-1: Predose | 0.0379 (0.392) | 0.00 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is 0. Below level of detection.
  MG-1: 0-2.5 h: number analyzed (Participants) | 105 | 25
  MG-1: 0-2.5 h | 12.0 (17.4) | 17.1 (37.4)
  MG-1: 2.5-5.0 h: number analyzed (Participants) | 98 | 17
  MG-1: 2.5-5.0 h | 12.0 (11.9) | 50.0 (67.1)
  MG-1:5.0-10 h: number analyzed (Participants) | 91 | 22
  MG-1:5.0-10 h | 8.51 (10.7) | 22.0 (21.4)
  MG-1: 8-24 h: number analyzed (Participants) | 71 | 11
  MG-1: 8-24 h | 3.25 (9.36) | 7.24 (10.1)
  MG-2: Predose | 0.0038 (0.039) | 0.00 (NA) — Mean of SUN13834 metabolite concentration at pre-dose is 0. Below level of detection.
  MG-2: 0-2.5 h: number analyzed (Participants) | 105 | 25
  MG-2: 0-2.5 h | 1.31 (2.84) | 1.78 (3.70)
  MG-2: 2.5-5.0 h: number analyzed (Participants) | 98 | 17
  MG-2: 2.5-5.0 h | 1.81 (3.58) | 6.98 (11.6)
  MG-2:5.0-10 h: number analyzed (Participants) | 91 | 22
  MG-2:5.0-10 h | 1.42 (3.40) | 4.93 (8.26)
  MG-2: 8-24 h: number analyzed (Participants) | 71 | 11
  MG-2: 8-24 h | 1.44 (3.57) | 1.60 (1.69)

19. Secondary Outcome: Summary of Treatment-Emergent Adverse Events in ≥2% of Participants Following Treatment With SUN13834 or Placebo in Adult Participants With Atopic Dermatitis
Description: Treatment-emergent adverse events (TEAEs) were defined as Adverse Events (AEs) that occurred from the time treatment was administered on Day 1 through the last follow-up visit or a worsening of a pre-existing condition.
Time Frame: Baseline up to Week 8 post-dose, up to a total of 36 weeks.
Population: Treatment-emergent adverse events were assessed using the Safety population. All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SUN13834 50 mg Tid | SUN13834 200 mg Tid
Number analyzed (Participants) | 120 | 120 | 30
Participants
  Number of participants with at least 1 Adverse Event | 82 | 68 | 14
  Bronchitis | 1 | 2 | 2
  Carbuncle | 0 | 0 | 1
  Influenza | 3 | 1 | 0
  Nasopharyngitis | 9 | 11 | 2
  Pneumonia | 0 | 0 | 1
  Sinusitis | 4 | 2 | 1
  Upper respiratory tract infection | 12 | 8 | 0
  Urinary tract infection | 0 | 1 | 2
  Diarrhea | 2 | 6 | 2
  Nausea | 5 | 6 | 0
  Vomiting | 3 | 0 | 1
  Blood creatine phosphokinase increased | 6 | 5 | 0
  Blood IgE increased | 0 | 1 | 1
  Blood pressure increased | 0 | 0 | 1
  Headache | 11 | 5 | 3
  Paresthesia | 0 | 0 | 1
  Dermatitis atopic | 3 | 2 | 1
  Pruritus | 2 | 2 | 1
  Rash | 0 | 0 | 1
  Oropharyngeal pain | 3 | 1 | 0
  Pulmonary Congestion | 0 | 0 | 1
  Fatigue | 0 | 0 | 1
  Joint injury | 0 | 1 | 1
  Pregnancy | 1 | 4 | 0
  Accelerated hypertension | 0 | 0 | 1
  Paranoia | 0 | 0 | 1
  Seasonal allergy | 0 | 1 | 1
  Cyst drainage | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) data were collected from Baseline (Day 1) up to 8 weeks post-dose, up to a total of 36 weeks.
Description: Treatment-emergent adverse events (TEAEs) were defined as Adverse Events (AEs) that occurred from the time treatment was administered on Day 1 through the last follow-up visit or a worsening of a pre-existing condition.
Groups:
- SUN13834 50 mg Tid: Participants with atopic dermatitis who were administered 2 SUN13834 tablets of 25 mg; 50 mg (2×25 mg) tid orally 3 times a day (tid) for 28 days.
- SUN13834 200 mg Tid: Participants with atopic dermatitis who were administered 2 SUN13834 tablets of 200 mg (2×100 mg) tid orally 3 times a day (tid) for 28 days.
Arm/Group | Placebo | SUN13834 50 mg Tid | SUN13834 200 mg Tid
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/120 | 0/120 | 0/30
Other Adverse Events (participants affected / at risk) | 46/120 | 44/120 | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | SUN13834 50 mg Tid (N=120) | SUN13834 200 mg Tid (N=30)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | SUN13834 50 mg Tid (N=120) | SUN13834 200 mg Tid (N=30)
Upper respiratory tract infection (Infections and infestations) | 12 | 8 | 0
Headache (Nervous system disorders) | 11 | 5 | 3
Nasopharyngitis (Infections and infestations) | 9 | 11 | 2
Blood creatine phosphokinase increased (Investigations) | 6 | 5 | 0
Nausea (Gastrointestinal disorders) | 5 | 6 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 6 | 2
Bronchitis (Infections and infestations) | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No